CLINICAL TRIAL: NCT00429780
Title: A Randomized, Safety, Immunogenicity & Efficacy Study of Autoclaved Leishmania Major Plus BCG vs. BCG (Double Blind) or Placebo (Open), in Healthy High Risk Iranian Volunteers With Positive Response to Leishmanin (LST>0)
Brief Title: Safety/Efficacy Trial of Killed Leishmania Vaccine in Volunteers With Positive Response to Leishmanin (LST>0)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Pasteur Institute of Iran, Tehran, Iran (Unknown); Razi Vaccine and Serum Research Institute (Other); Centre for Disease Control & Management, Ministry of Health & Medical Education (Other Government)
Responsible Party: Ali Khamesipour, Center for Research & Training in Skin Diseases & Leprosy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J/423/1058, 30/05/1385
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Leishmaniasis vaccine; Alum-ALM; First generation vaccine; Leishmanin positive; Healthy Volunteers; Response to Leishmanin (Leishmanin Skin Test>0); No History of Cutaneous Leishmaniasis

ARMS (2):
- Alum-ALM + BCG (No Intervention): Alum-ALM + BCG
- Placebo (No Intervention): BCG diluent
  Interventions: Biological: Alum-ALM + BCG

INTERVENTIONS:
Biological: Alum-ALM + BCG — Alum-ALM + BCG 200 ug per injection
  Other Names: Alum pericipitated autoclaved L. major
  Arms: Placebo

SUMMARY:
Development of a safe and effective vaccine against leishmaniasis started more than 10 years ago under WHO/TDR supervision. An autoclaved L. major vaccine (ALM) mixed with BCG has been tested in human in Iran, Pakistan and Sudan. Long term follow up of the vaccinees showed no untoward reactions except the skin reaction at the site of injection. The efficacy results of ALM was not satisfactory. In order to enhance immunogenicity of the vaccine, ALM was adsorbed to alum (Aluminum hydroxide). Alum-ALM plus adjuvant showed to induce protection in Rhesus monkeys against cutaneous leishmaniasis and in Languor monkeys against visceral leishmaniasis. Two trials of a single injection of different doses of Alum-ALM mixed with 1/10th of normal dose of BCG was carried out in healthy volunteers from a non endemic area of Sudan. The safety/immunogenicity parameters of the volunteers were closely monitored and the results showed that side effects were minimal and confined to the site of injection in the form of mild local pain, induration and ulceration, all associated with BCG vaccination. The immunogenicity results showed the strongest immune response seen in any Leishmania vaccine trials so far. It seems that this new formulation is an appropriate candidate for further development. Inoculation with live virulent Leishmania to produce a lesion for the purpose of preventing natural infection is known as leishmanization. The induced lesion heals and the person is usually protected against further infections. This method of prevention was practiced for centuries in the region. In this study volunteers with response to leishmanin will be injected twice (30 days apart) with Alum-ALM 200 ug + 1/10 of BCG (n = 50) or diluent alone (n = 50) as control. All volunteers will be leishmanized on day 60 post vaccination. In this trial, volunteers are protected either by vaccine or by leishmanization. The leishmanized volunteers will be visited by weekly and the development and healing process of the lesion will be monitored until complete healing of every volunteer. The immune responses of the volunteers will be evaluated. Vaccine efficacy is defined by the percent reduction in the number of volunteers developing a lesion following leishmanization as compared to controls on days 240.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age between 16 to 60 years.
* Generally in good health.
* No known immunological deficiency, including HIV infection (by medical history).
* No fever at the time of vaccination i.e. oral body temperature <37.5°C.
* No history/suspicion/presence of kala-azar or cutaneous leishmaniasis (CL).
* No history of leishmanization.
* No history of vaccination against leishmaniasis.
* No involvement in other drug or vaccine trial(s) during the study period.
* No other known or planned vaccination within 1 month prior to the study and during the study period.
* No current or foreseeable use of immunosuppressors (i.e. corticosteroids) within one month prior to the vaccination and during the period of the study.
* No known allergy to a vaccine component (e.g. BCG, alum hydroxide, etc.).
* Written informed consent provided. If the volunteer is under 18 years old, the legal guardian's signature is required on the informed consent.

Exclusion Criteria:

* Pregnancy.
* Women should not be pregnant and/or lactating and/or planning pregnancy throughout the study period until complete healing of the lesion induced by vaccination and/or leishmanization.
* A urinary pregnancy test will be performed for all women of child bearing potential at entry and adequate contraception throughout the study should be used if applicable.
* Evidence of prior CL or leishmaniasis (e.g. sign of scar resembling leishmaniasis, confirmed by physical examination).
* Evidence of serious diseases, allergy or allergic conditions leading to medical consultation and treatment especially with steroids or levamisole, recent surgery or hospitalisation, according to the physical examination and medical history interview.
* Presence of any chronic illness/disease including diabetes mellitus, tuberculosis, leprosy, epilepsy and hypertension.
* Abnormal haematology and clinical chemistry (See Sections 8.1.2.1 and 8.1.2.2 for normal ranges of laboratory values).
* Presence of fever at the time of vaccination, i.e. body temperature (by mouth) > 37.5°C.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of local/systemic adverse events after vaccination assessed by
interview, physical examination in volunteers with a response to
Leishmanin (LST>0);
Percentage of the volunteers with LST>0 protected against CL
(absence of a lesion).

SECONDARY OUTCOMES:
Percentage of volunteers partially protected against CL compared to controls at day 240.
To assess immune response of the volunteers at baseline (prior to vaccination), before leishmanization to evaluate the immunogenicity of the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khamesipour, Principal Investigator — Center for Research and Training in Skin Disease and Leprosy,
Locations (1):
- Center for Research & Training in Skin Diseases & Leprosy, Tehran, Iran